CLINICAL TRIAL: NCT03716921
Title: Short 3-week Antibiotic Treatment Versus 6 Weeks in Adults With Septic Arthritis of Native Joint: a Randomized, Open Label, Non-inferiority Trial
Brief Title: Short 3-week Antibiotic Treatment Versus 6 Weeks in Adults With Septic Arthritis of Native Joint
Acronym: SHASAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P170911J; IDRCB (Other: 2018 - A02040-55)
Record Dates: First submitted 2018-10-10; First posted 2018-10-23 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Septic Arthritis
Keywords: Septic Arthritis of native joint; short antibiotic treatment; native joint; septic arthritis
MeSH Terms: conditions — Arthritis, Infectious

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short antibiotics treatment (Experimental): patients will receive effective antibiotic treatment (IV and oral) for 3 weeks
  Interventions: Other: Short antibiotics treatment
- Long antibiotics treatment (No Intervention): patients will receive effective antibiotic treatment (IV and oral) for 6 weeks according to standard care

INTERVENTIONS:
Other: Short antibiotics treatment — Patients randomized in this arm will pursue antibiotic administration until visit 3 weeks after D0
  Other Names: 3-week antibiotic treatment
  Arms: Short antibiotics treatment

SUMMARY:
In France, the incidence of native joint infections is about 10 per 100 000 person-years, most commonly caused by S.aureus followed by b-haemolytic streptococci. French and international antibiotic guidelines, based on expert advice and retrospective studies, recommend intravenous antibiotics for two weeks, then oral for 4 weeks without evident link between intravenous, prolonged oral treatment and cure. Long term exposure to antibiotics increases bacterial resistance, a major problem of public health. Several studies show that serious infectious can be treated safely by a shorter treatment and with oral antibiotics. There is no randomized controlled trial to establish the duration of antibiotics in native joint infections. Moreover, no consensus prevails on the administration route and duration of antimicrobial therapy. Although most clinicians acknowledge the interest of oral antibiotics and shorter treatment duration, randomized controlled trials are necessary to evaluate this practice. The SHASAR project aims to evaluate whether a shorter antibiotic treatment (3 week treatment) is safe and not inferior to the conventional 6 week treatment in native joint infections. If successful, this would represent a major advance in terms of patients' quality of life; decreased rate of health-care-related infections and complications, bacterial resistance and cost.

DETAILED DESCRIPTION:
This trial is a nationwide, non inferiority, multicenter French randomized, open-label, controlled trial comparing two treatment durations, 3 versus 6 weeks, in septic arthritis of native joints. Patients who fulfill inclusion criteria will be randomized between day0 and day5. Day 0 is the time when effective intravenous antibiotic treatment is started. Effective treatment is defined by active antibiotics on the identified bacteria according to the susceptibility. The randomisation (1:1 ratio) will be stratified on early planned drainage. Follow-up will include 6 visits and will consist in clinical, biological, radiological, health quality of life (EQ-5D-3L score) and adverse events record. After collection, validation of data and population description, analysis will be conducted on the per-protocol population (patients receiving the planned duration of antibiotic +/-3days). This study will not be carried out blind for feasibility reasons. According to statistical considerations (by accounting for 5% of subjects lost to follow-up), the required sample size will be of 350 patients overall.

ELIGIBILITY:
Inclusion Criteria:

* Septic arthritis of native joint defined by: 1) clinical signs (hot and/or swollen and/or tender and painful joint (measured by a visual analogue scale)) and 2) microbiologically confirmed pyogenic arthritis (microorganism cultured in the synovial fluid joint or in the blood with complete bacterial susceptibility)
* Patients aged of 18 years or older
* Informed, written consent obtained from the patient
* Patient having the rights to French social insurance

Exclusion Criteria:

* Prosthetic joints
* Septic arthritis in the past 12 months
* Osteomyelitis
* Diabetic foot
* Septic choc
* Arthritis due to bacteria resistant to available oral antibiotics
* Arthritis due to the following microorganisms: Mycobacterium, fungi, Brucella, Borrelia, Neisseria gonorrhoeae, Neisseria meningitidis, Nocardia, Mycoplasma spp, Pseudomonas aeruginosa.
* Glomerular filtration rate < 30ml/min/1,73m2
* Neutrophils < 500/mm3
* Difficulties regarding compliance with oral antibiotics
* Contraindication to oral antibiotics necessary to treat joint infection
* Pregnancy or lactating woman
* Curator or guardianship
* Participation in other interventional research during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Cure at 16 weeks (4 months) after the beginning of the treatment | 16 weeks after Day 0
  Cure is defined as absence of clinical signs of joint infection, absence of treatment failure, absence of relapse

SECONDARY OUTCOMES:
Cure at 24 weeks | 24 weeks after Day 0
  Cure is defined as absence of clinical signs of joint infection, absence of treatment failure, absence of relapse
Treatment failure and relapse and relapse rates | 6,16,24 weeks after Day 0
  % of relapse at 6,16,24 weeks
The patient's quality of life | 3,6,16,24 weeks after Day 0
  assessed by a quality of life questionnaire on 3,6,16,24 weeks. The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
The residual joint pain in the affected joint | at 16 and 24 weeks after Day 0
  The residual joint pain is measured by a numerical scale. 0 means "no pain at all" and 10 "pain as bad as it could be".
hospital length of stay and total treatments costs | through study completion, an average of 3 years
  To compare cost-effectiveness and cost utility of 3-week vs 6-week antibiotic strategies for patients with arthritis of native joints
joint mobility | at 16 and 24 weeks after Day 0
  joint mobility is assessed by "good mobility, few mobility, no mobility"

CONTACTS AND LOCATIONS:
Overall Officials: Lélia ESCAUT, Dr, Principal Investigator — AP-HP Hôpital Bicêtre
Locations (31):
- France (31):
  - Hôpital Avicenne - Service de Rhumatologie, Bobigny
  - Hôpital Pellegrin Bordeaux - Service de Rhumatologie, Bordeaux
  - Hôpital Ambroise Paré - Service de Rhumatologie, Boulogne-Billancourt
  - Hôpital Cavale Blanche - Service de Maladies Infectieuses, Brest
  - CHG Pontoise - Centre Hospitalier René Dubos - Service de Rhumatologie, Cergy-Pontoise
  - CHU Tours - Hôpital Trousseau - Service de Rhumatologie, Chambray-lès-Tours
  - Hôpital Antoine Béclère - Service de Maladies Infectieuses, Clamart
  - CHSF - Service de Rhumatologie, Corbeil-Essonnes
  - CHU Dijon Bourgogne - Hôpital François Mitterrand -Service de Maladies Infectieuses, Dijon
  - CHU Grenoble Alpes - Hôpital Sud - Service de Rhumatologie, Échirolles
  - Hôpital Raymond Poincaré - Service de Maladies Infectieuses, Garches
  - CHU Grenoble Alpes - Hôpital Michallon - Service de Maladies Infectieuses, La Tronche
  - Hopital Bicêtre, Service de Maladies Infectieuses et Tropicales, Le Kremlin-Bicêtre
  - Hôpital Bicêtre service de rhumatologie, Le Kremlin-Bicêtre
  - CHRU Lille - Service de Rhumatologie, Lille
  - CHR Orléans - Service de Rhumatologie, Orléans
  - Hôpital Lariboisière Service de Rhumatologie, Paris
  - Hôpital Saint Antoine - Service de Rhumatologie, Paris
  - Hôpital Pitié Salpetrière - Service de Maladies Infectieuses, Paris
  - Hôpital Pitié Salpetrière - Service de Rhumatologie, Paris
  - Hôpital Cochin - Service de Maladies Infectieuses, Paris
  - Hôpital Cochin - Service de Rhumatologie, Paris
  - Hôpital Bichat - Service de Rhumatologie, Paris
  - GH Diaconesse La Croix St Simon - Service de Rhumatologie, Paris
  - Hôpital Sud Rennes - Service de Rhumatologie, Rennes
  - CHU Saint Etienne - Hôpital Nord - Service de Maladies Infectieuses, Saint-Priest-en-Jarez
  - CHU Saint Etienne - Hôpital Nord - Service de Rhumatologie, Saint-Priest-en-Jarez
  - CHRU Strasbourg - Hôpital de Hautepierre - Service de Rhumatologie, Strasbourg
  - CHU Tours - Hôpital Bretonneau - Service de Maladies Infectieuses, Tours
  - Hôpitaux de Brabois - Service de Maladies Infectieuses, Vandœuvre-lès-Nancy
  - Hôpitaux de Brabois - Service de Rhumatologie, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No